CLINICAL TRIAL: NCT01553643
Title: A Randomized Double Blind Placebo Control Study of Huang-Chi-Wu-Wu- Tang in Patients With Intracranial Arterial Stenosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DMR98-IRB-281
Record Dates: First submitted 2012-03-07; First posted 2012-03-14 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2012-03

CONDITIONS: Intracranial Arterial Stenosis
Keywords: Huang-Chi-Wu-Wu-Tang; Intracranial arterial prominent stenosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Chinese Herb Huang-Chi-Wu-Wu-Tang (Experimental)
  Interventions: Drug: Chinese Herb Huang-Chi-Wu-Wu-Tang
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Chinese Herb Huang-Chi-Wu-Wu-Tang — Huang-Chi-Wu-Wu-Tang at a rate of 3g two times per day
  Arms: Chinese Herb Huang-Chi-Wu-Wu-Tang
Drug: placebo — at a rate of 3g two times per day
  Arms: Placebo

SUMMARY:
Intracranial arterial prominent stenosis (IAPS) is one of main cause of stroke especially in Asia. Although antiplatelet aggregative or anticoagulant agent and even surgical operation are used to treat patients with IAPS, the incidence of stroke occurrence still remains high. In addition, symptomatic IAPS most common cause continuous deterioration, thus, increase the incidence of stroke. Therefore, there is a good method to reduce the inceidence of stroke that is to prevent the progressive deterioration of IAPS.

Huang-Chi-Wu-Wu-Tang is made of Astrgalus membranaceus (Fisch.) Gge , Paeonia lactiflora Pall , Cinnamom Twig , Zingiber officinale Rose , Ziziphus jujube Mill , and can treat hemiplegia in the traditional Chinese medicine writings. Astragaloside IV is a component of Astrgalus membranaceus, may reduce th cerebral infarction area in middle cerebral arterial occlusion mice. The investigators previous studies have known that paeoniflorin that a component of Paeonia lactiflora Pall can decrease the cerebral infarction area and neurological deficit in middle cerebral arterial occlusion rats. Therefore, the purpose of the present study was to investigate the effect of Huang-Chi-Wu-Wu-Tang on patients with IAPS.

ELIGIBILITY:
Inclusion Criteria:

1. Had received Transcranial Doppolar Sonography.
2. Age >40 years old.
3. Gender: Male or female.
4. The subject or their legal representative gave written informed consent to participate.
5. Meet with one of the two Transcranial Doppolar Sonography results below:

   * The evaluated standard of MCA M1 stenosis of 50-99% are as follows:

     * PSV >140 cm/s
     * MFV >100 cm/s
   * The evaluated standard of BA stenosis of 50-99% are as follows:

     * PSV >100 cm/s
     * MFV >60 cm/s

Exclusion Criteria:

1. Refused to sign the Informed Consent Form.
2. Too irritable to accept the evaluation.
3. Age ≦40 years old.
4. Major diseases such as Myocardial Infarction、Heart failure、Chronic pulmonary obstructive disease(COPD）with dyspnea、Liver failure or Renal failure.
5. Pregnancy or breast-feeding.

Min Age: 41 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-01; Primary Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Primary outcome measure was the improvement hemodynamics at intracranial vessels in the M1 segment of middle cerebral artery (MCA) or basilar artery (BA) shown in transcranial color-coded sonography (TCCS). | 3 years(all patients)

CONTACTS AND LOCATIONS:
Overall Officials: Chung Hsiang Liu, MD., Principal Investigator — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taiching, Taiwan